CLINICAL TRIAL: NCT02897947
Title: Outcome of Surgery for Lumbar Spinal Stenosis - a Comparison of Data From Three National Quality Registries
Status: Completed | Type: Observational
Sponsor: St. Olavs Hospital (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Sponsor
Other Study IDs: 2014/2219
Record Dates: First submitted 2016-09-07; First posted 2016-09-13 (Estimated); Last update posted 2018-09-05 (Actual); Status verified 2018-08

CONDITIONS: Spinal Stenosis; Intermittent Claudication
Keywords: Lumbosacral Region; Surgery; Registries
MeSH Terms: conditions — Spinal Stenosis; Intermittent Claudication | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- treated in Norway included in NORspine: patients having had surgery for lumbar spinal stenosis in Norway and are included in the national register NORspine
  Interventions: Procedure: Surgery for lumbar spinal stenosis in Norway
- treated in Sweden included in Swespine: patients having had surgery for lumbar spinal stenosis in Sweden and are included in the national register Swespine
  Interventions: Procedure: Surgery for lumbar spinal stenosis in Sweden
- treated in Denmark included in Danespine: patients having had surgery for lumbar spinal stenosis in Denmark and are included in the national register DANEspine
  Interventions: Procedure: Surgery for lumbar spinal stenosis in Denmark

INTERVENTIONS:
Procedure: Surgery for lumbar spinal stenosis in Norway
  Other Names: Surgery for neurogenic claudication due to lumbar spinal stenosis in Norway
  Groups: treated in Norway included in NORspine
Procedure: Surgery for lumbar spinal stenosis in Sweden — Surgery for neurogenic claudication due to lumbar spinal stenosis in Sweden
  Groups: treated in Sweden included in Swespine
Procedure: Surgery for lumbar spinal stenosis in Denmark — Surgery for neurogenic claudication due to lumbar spinal stenosis in Denmark
  Groups: treated in Denmark included in Danespine

SUMMARY:
There is no international consensus on evaluation and surgical treatment of Lumbar Spinal Stenosis (LSS). The indication for operative treatment is relative, and the variation in surgical rates and procedures is significant, both within and between countries. Understanding practice-based variety is critical since these differences may reflect a disparity in quality of the health care in different institutions, regions, or countries. Norway, Sweden, and Denmark do all have National spine registers for research and quality assessment. Comparing indications for surgery, selected procedure, patient reported outcomes, and factors predicting outcome after surgery for LSS between these countries could provide information about optimal indications and strategy for surgery. Register-based studies have advantages such as large sample sizes and high external validity, but also limitations such as lower follow-up rates, and inferior data quality compared to clinical trials.

Hypotheses: Between these three countries, there are no differences in (i) indications for surgery, (ii) patient-reported outcome after surgery or (iii) risk factors associated to outcome are similar.

DETAILED DESCRIPTION:
This is an observational register based study, i.e. prospective data registration and a retrospective study design. Eligible patients are those 50 years or older treated surgically for LSS in Denmark, Norway or Sweden during 2011, 2012, or 2013 with no history of previous lumbar spine surgery. Register-based studies have advantages such as large sample sizes and greater external validity, but also limitations such as lower follow-up rates, inferior data quality compared to clinical trials. Data will be presented according to the STROBE criteria.

The registers:

All registries have the aim of studying outcome after spine surgery. All departments participate voluntarily. Patients participate voluntarily after signing an informed consent. At the time of admission, the patient reports data on demographics, social factors, comorbidity and previous surgery. After surgery, the surgeon records diagnosis and type of surgery performed.

The Norwegian Spine register, NORspine, is based on experiences from the Swespine register and previous validation studies from a local clinical registry, and was founded in 2007. In total 38 of 40 centers performing lumbar spine surgery in Norway report to NORspine. Coverage is approximately 95%. The completeness is approximately 65%.

The Swespine Register has included individuals treated with surgery for lumbar spinal stenosis since 1993. During the last decade, the number of departments participating in the registry has varied between 35 and 41 of the 42 to 45 departments providing spinal surgery services in Sweden. Coverage is approximately 90%. The completeness (number of patients reported to Swespine at the time of surgery) is approximately 80%.

The Danish spine register, DaneSpine, is based on Swespine and was acquired by the Danish Spine Society from the Swedish Society of Spinal Surgeons in 2009 and has successively been implemented. Coverage and completeness for DaneSpine has not been determined.

Quality assurance:

Loss to follow-up may bias the results. Solberg et al. (2011) studied 633 patients, who were operated on for degenerative disorders of the lumbar spine in Norway, and found that a loss to follow-up of 22% would not bias conclusions about overall treatment effects. There were no indications of worse outcomes in the non-responders group. In a similar one-center study of the DaneSpine. Højmark et al. (2016) found that a loss to follow-up of 12% at did not seem to bias the conclusions that can be drawn from DaneSpine at that center.

Data handling Anonymized individual level data from all three registers will be pooled in one database. The cohort will be divided by country for comparisons.

Missing data and out of range data: In case of missing data case exclusion analysis by analysis, will be used. Out of range data will be deleted.

Analysis The data will be cleaned by excluding patients with missing or incorrect date of surgery, missing date for follow-up, previous lumbar spine surgery and surgery other than decompression for lumbar spinal stenosis with or without concomitant arthrodesis.

After data cleaning, we aim to perform blinded statistical analyses, in which the independent statistician performing the analyses is unaware of group belonging (i.e. country). The code will not be broken until the analyses and interpretations have been performed.

Comparisons of indications for surgery Analysis of baseline data will include age at surgery, sex, anthropometrics, number of smokers, Oswestry Disability Index, EQ-5D, number on sick leave, employment status, and duration of leg and back pain and presented as mean (SD), mean (95% confidence interval), or number (%).

Variables will be analyzed by analysis of variance, Chi-square or logistic regression tests. Data will be presented as crude (unadjusted) data to elucidate any differences between the countries.

Comparisons of outcome Comparisons of the change of the outcome variables from baseline to 1 year, as well as comparisons of the actual value at 1 year will be performed. Analysis of covariance, Chi-square or logistic regression tests and the crude (unadjusted) data will be presented.

In addition, baseline variables will be used as covariates in the analysis of covariance and the adjusted data presented. Propensity scores will also be considered as covariates.

Comparison of surgical method used Based on the decompression with or without concomitant arthrodesis. Non-response analysis A non-response analysis will be performed comparing all available baseline variables between those that responded to the 1 year follow-up with those that did not respond.

Sample size A study of similar character has never been performed before. Due to the nature of the study, the sample size is not formulated in the guise of power, risk level, or clinical difference. The number of patients participating in the study is estimated to 7500. The sample is so large that differences in the Oswestry Disability Index of as low as 2 points may be detected (power 90%, significance level 5%), but in the interpretation the minimal important difference of 10-15 points in the Oswestry Disability Index often referred to has to be taken into account.

ELIGIBILITY:
Inclusion Criteria:

* treated with surgery for lumbar spinal stenosis in Norway, Sweden or Denmark
* registered in a national quality register
* signed informed consent

Exclusion Criteria:

* not treated with decompression with or without concomitant arthrodesis for the lumbar spinal stenosis

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals treated surgically for lumbar spinal stenosis in Denmark, Norway and Sweden during 2011, 2012 and 2013 are included.
Sampling Method: Non-Probability Sample
Enrollment: 7500 (Actual)
Dates: Start 2011-01; Primary Completion 2013-12 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Oswestry disability index version 2.1 | preoperative and 1 year postoperative
  (from 0; no disability to 100; maximum disability) Index at baseline, index change from preoperative to 1year follow-up and actual index at 1 year follow-up.

SECONDARY OUTCOMES:
Numerical rating scale for leg pain (from 0; no pain to 10; maximum pain) | preoperative and 1 year postoperative
  The numerical rating scale is used in Norway. The visual analogue scale (0-100) used in Sweden and Denmark will be converted to the numerical rating scale. Index at baseline, index change from preoperative to 1 year follow-up and actual index at 1 year follow-up
Numerical rating scale for back pain (from 0; no pain to 10; maximum pain) | preoperative and 1 year postoperative
  The numerical rating scale is used in Norway. The visual analogue scale (0-100) used in Sweden and Denmark will be converted to the numerical rating scale. Index at baseline, index change from preoperative to 1-year follow-up and actual index at 1 year follow-up.
European Quality of Life-5 Dimensions (EQ-5D) according to the British tariff (UK-time tradeoff, TTO); from -0.59; worst possible health to 1; perfect health) | preoperative and 1 year postoperative
  Index at baseline; change from preoperative to 1-year follow-up and actual index at 1-year follow-up.
Return to work rate | preoperative and 1 year postoperative
Operation method: Decompression with or without concomitant arthrodesis for the lumbar spinal stenosis. | preoperative
Additional surgery in the lumbar spine | during 1 year follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Greger Lønne, md phd, Principal Investigator — St. Olavs Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lonne G, Fritzell P, Hagg O, Nordvall D, Gerdhem P, Lagerback T, Andersen M, Eiskjaer S, Gehrchen M, Jacobs W, van Hooff ML, Solberg TK. Lumbar spinal stenosis: comparison of surgical practice variation and clinical outcome in three national spine registries. Spine J. 2019 Jan;19(1):41-49. doi: 10.1016/j.spinee.2018.05.028. Epub 2018 May 21. PMID 29792994